CLINICAL TRIAL: NCT03670992
Title: Case Series: Combined, Surgical-only Treatment of Pancreatic and Extra-pancreatic Metastases From Renal Cell Carcinoma - a Quality of Life and Survival Analysis
Brief Title: Surgical Treatment of Pancreatic RCC Metastases
Status: Completed | Type: Observational
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Professor Stefania Brozzetti, Professor, Azienda Policlinico Umberto I
Other Study IDs: PAN001
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Renal Cell Carcinoma; Metastases, Neoplasm
Keywords: renal cell carcinoma; pancreatic resection; robotic surgery; pancreatic metastases; quality of life
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic Metastases: Patients with only pancreatic metastases from RCC
  Interventions: Procedure: duodenal-pancreatectomy
- extra-pancreatic metastases: patients with extra pancreatic metastases from RCC
  Interventions: Procedure: duodenal-pancreatectomy

INTERVENTIONS:
Procedure: duodenal-pancreatectomy — surgical removal of metastatic repetitions in pancreas and/or other distal sites
  Other Names: total-pancreatectomy; distal-pancreatectomy; other metastases resection

SUMMARY:
Data from 26 patients undergoing resection of Pancreatic Metastases and extra-Pancreatic Metastases from RCC were retrospectively analysed. Clinical data were collected from a digital database and QoL was assessed through patient's interview and Karnofsky performance scale.

DETAILED DESCRIPTION:
Retrospective data was analysed from 26 patients that were submitted to pancreatic resection between August 2002 and November 2015. Inclusion criteria were: single or multiple metastases in pancreas or extra pancreatic; primary RCC; never received chemotherapic treatment; patients that already received a previous pancreatic resection were also included.

Cases were collected from two high-volume centres: Surgical Department "Pietro Valdoni" in Policlinico Umberto I and the Division of Transplantation and General Surgery at University of Pisa.

Different kind of surgical approaches were taken into account in this study: duodenal-pancreatectomy, total-pancreatectomy and distal-pancreatectomy associated or not with other metastatic site resections. Surgery was performed either with classical open approach and modern robotic surgical approach, with the robot "Da Vinci". Aim of surgical interventions were to remove all metastases in association to radical lymphadenectomy thus to achieve R0 result. All postoperative events occurring within 90 days of surgery were considered. Postoperative complications were graded according to Clavien-Dindo classification.

Patients were followed-up 3 months after discharge and every 6 months thereafter.

Patients had blood chemistries and CT scans at least every year. A database was used to record all patients' data. Results were analysed in terms of Operative Mortality and Morbidity, Actuarial Survival, Actuarial Disease-Free Survival and Quality of Life.

Protocols were approved by the bioethical review committee and meet the guidelines of both University Sapienza of Rome and University of Pisa.

QoL was measured by Karnofsky performance scale and through Activities of Daily Living scale (ADL), Instrumental Activities of Daily living scale (IADL), BMI evaluation, serum albumin and hemoglobin, also depression was evaluated as a parameter. QoL was defined by combination of these parameters as: excellent, good, fair, poor or very poor.

A low Karnofsky scale index with inadequate social and environmental situations, a reduction in functional capacity with depression and severe weight-loss were identified as a decline in QoL.

Data was analysed via Chi-square test, as well as Student's paired and unpaired t-tests.

Actuarial relative survival and actuarial relative disease-free survival were described by Kaplan-Meier analysis. A log-rank test was used to compare continuous variables and was expressed by Kaplan-Meier curves. Homogeneity of the different groups to be compared was tested by chi-square test. Statistical significance was set at p ≤ 0,05.

ELIGIBILITY:
Inclusion Criteria:

* metastases from RCC
* surgically manageable lesions

Exclusion Criteria:

* metastases from different malignancies
* other malignancies
* surgically unmanageable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 26 patients, 12 male and 14 female age range 46 - 83, mean age 66 SD 9,1
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Survival | follow up 36 months
  Three years survival
Survival 2 | follow up 60 months
  five years survival
Survival 3 | follow up 120 months
  ten years Survival

SECONDARY OUTCOMES:
Karnofsky scale | mean follow up 45 months range (6-163 months)
  common scale to evaluate patient's prognosis in clinical and surgical settings. Adimensional scale in a range of 0-100. Higher Karnofsky score is associated with better outcome, score is assessed in steps of 10 (0 - 10 - 20 - 30 - 40 - 50 - 60 - 70 - 80 - 90 - 100).
Activity of daily living scale (ADL scale) | mean follow up 45 months range (6-163 months)
  prognostic scale evaluated through validated questionnaires, adimensional scale in a range of 0-6 points. evaluates abilty of the patients to fullfill the common daily activities. Better outcome is associated with higher score.
Instrumental Activity of daily living scale (IADL scale) | mean follow up 45 months range (6-163 months)
  prognostic scale evaluated through validated questionnaires, adimensional scale in a range of 0-8 points. Evaluates ability of the patient to use the common day instruments. Better outcome is associated with higher score.
Nutritional status | mean follow up 45 months range (6-163 months)
  BMI monitoring in kg/m^2
Serum albumin | mean follow up 45 months range (6-163 months)
  Serum albumin monitoring in g/dl
Hemoglobin | mean follow up 45 months range (6-163 months)
  Hemoglobin monitoring in g/dl

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Brozzetti, professor, Study Director — Policlinico Umberto I
Locations (1):
- Department of Surgery "Pietro Valdoni", Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adler H, Redmond CE, Heneghan HM, Swan N, Maguire D, Traynor O, Hoti E, Geoghegan JG, Conlon KC. Pancreatectomy for metastatic disease: a systematic review. Eur J Surg Oncol. 2014 Apr;40(4):379-86. doi: 10.1016/j.ejso.2013.12.022. Epub 2014 Jan 15. PMID 24462547
- [Result] Tanis PJ, van der Gaag NA, Busch OR, van Gulik TM, Gouma DJ. Systematic review of pancreatic surgery for metastatic renal cell carcinoma. Br J Surg. 2009 Jun;96(6):579-92. doi: 10.1002/bjs.6606. PMID 19434703
- [Result] Grassi P, Doucet L, Giglione P, Grunwald V, Melichar B, Galli L, De Giorgi U, Sabbatini R, Ortega C, Santoni M, Bamias A, Verzoni E, Derosa L, Studentova H, Pacifici M, Coppa J, Mazzaferro V, de Braud F, Porta C, Escudier B, Procopio G. Clinical Impact of Pancreatic Metastases from Renal Cell Carcinoma: A Multicenter Retrospective Analysis. PLoS One. 2016 Apr 11;11(4):e0151662. doi: 10.1371/journal.pone.0151662. eCollection 2016. PMID 27064898
- [Result] Fikatas P, Klein F, Andreou A, Schmuck RB, Pratschke J, Bahra M. Long-term Survival After Surgical Treatment of Renal Cell Carcinoma Metastasis Within the Pancreas. Anticancer Res. 2016 Aug;36(8):4273-8. PMID 27466543
- [Derived] Brozzetti S, Bini S, De Lio N, Lombardo C, Boggi U. Surgical-only treatment of pancreatic and extra-pancreatic metastases from renal cell carcinoma - quality of life and survival analysis. BMC Surg. 2020 May 13;20(1):101. doi: 10.1186/s12893-020-00757-0. PMID 32404091